CLINICAL TRIAL: NCT00012038
Title: A Phase I/II Trial Of MGI114 For Treatment Of Patients With Recurrent Malignant Gliomas
Brief Title: Chemotherapy in Treating Patients With Progressive or Recurrent Brain Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New Approaches to Brain Tumor Therapy Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068474; NABTT-2005; JHOC-NABTT-2005
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2003-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Gliosarcoma | interventions — irofulven

INTERVENTIONS:
Drug: irofulven

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of irofulven in treating patients who have progressive or recurrent astrocytoma, oligodendroglioma, or glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of irofulven alone or combined with anticonvulsants known to be metabolized by cytochrome P450 in patients with progressive or recurrent high-grade anaplastic astrocytoma, anaplastic oligodendroglioma, or glioblastoma multiforme.
* Assess the pharmacokinetics of this drug on this schedule and determine the effects of P450-inducing anticonvulsants on the pharmacokinetics in these patients.
* Determine the response rate of patients treated with this drug administered at the MTD.
* Determine the duration of progression-free survival and overall survival of patients treated with this drug.
* Determine the toxic effects of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to concurrent use of anticonvulsant drugs that induce cytochrome P450 (yes vs no drugs or modest-induction drugs).

Patients receive irofulven IV over 30 minutes on days 1-4 or 1-5 (depending on dose-escalation level). Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients (per stratum) receive escalating doses of irofulven until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued to receive treatment with irofulven at the recommended phase II dose.

Patients are followed at 1 week and then every 2 months thereafter.

PROJECTED ACCRUAL: Approximately 18 patients (9 per stratum) will be accrued for the phase I portion of the study. Approximately 17-35 patients will be accrued for the phase II portion of the study within 6-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven malignant high-grade glioma that is progressive or recurrent after radiotherapy and/or chemotherapy

  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Glioblastoma multiforme
* Prior low-grade glioma that has progressed to high-grade glioma after radiotherapy and/or chemotherapy allowed
* Measurable disease by MRI or CT scan

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* Transaminases no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious concurrent infection or medical illness that would preclude study therapy
* No other prior malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast
* Mini mental score at least 15

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No more than 2 prior chemotherapy regimens
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered

Endocrine therapy:

* Maintained on a stable corticosteroid regimen for at least 5 days before and during study

Radiotherapy:

* See Disease Characteristics
* At least 3 months since prior radiotherapy and recovered

Surgery:

* Recovered from prior surgery

Other:

* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07; Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven S. Rosenfeld, MD, PhD, Study Chair — University of Alabama at Birmingham
Locations (10):
- United States (10):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas